CLINICAL TRIAL: NCT02447497
Title: Assessment of Antimicrobial Persistence of 3M CHG/IPA Preoperative Skin Preparation Against Resident Flora on the Abdominal and Inguinal Regions
Brief Title: In Vivo Patient Preoperative Skin Prep Persistence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Solventum US LLC (Industry)
Collaborators: 3M (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: EM-05-013509
Record Dates: First submitted 2015-05-08; First posted 2015-05-19 (Estimated); Results first posted 2020-11-23 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: Bacterial Recovery of Skin Flora Post-Product Application

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- 3M CHG/IPA - Abdominal Region (Experimental): Apply Chlorhexidine (CHG) 2% / Isopropyl alcohol (IPA) 70% for 30 seconds and allow to dry for 3 minutes.
  Interventions: Drug: 3M CHG/IPA Surgical Skin Preparation - Abdominal Region
- Normal Saline - Abdominal Region (Placebo Comparator): Apply 0.9% sodium chloride with applicator for 30 seconds and allow to dry for 3 minutes.
  Interventions: Other: Normal Saline - Abdominal Region
- 3M CHG/IPA - Inguinal Region (Experimental): Apply Chlorhexidine (CHG) 2% / Isopropyl alcohol (IPA) 70% for 30 seconds and allow to dry for 3 minutes.
  Interventions: Drug: 3M CHG/IPA Surgical Skin Preparation - Inguinal Region
- Normal Saline - Inguinal Region (Placebo Comparator): Apply 0.9% sodium chloride with applicator for 30 seconds and allow to dry for 3 minutes.
  Interventions: Other: Normal Saline - Inguinal Region

INTERVENTIONS:
Drug: 3M CHG/IPA Surgical Skin Preparation - Abdominal Region — Chlorhexidine gluconate 2% / Isopropyl alcohol 70%
  Other Names: SoluPrep
  Arms: 3M CHG/IPA - Abdominal Region
Other: Normal Saline - Abdominal Region — 0.9% sodium chloride applied with foam applicator
  Arms: Normal Saline - Abdominal Region
Drug: 3M CHG/IPA Surgical Skin Preparation - Inguinal Region — Chlorhexidine gluconate 2% / Isopropyl alcohol 70%
  Other Names: SoluPrep
  Arms: 3M CHG/IPA - Inguinal Region
Other: Normal Saline - Inguinal Region — 0.9% sodium chloride applied with foam applicator
  Arms: Normal Saline - Inguinal Region

SUMMARY:
The objective of the study is to demonstrate persistence of the CHG/IPA Prep on skin flora of the abdominal and inguinal regions of human subjects.

DETAILED DESCRIPTION:
The objective of the study is to demonstrate persistence of the CHG/IPA Prep versus a saline placebo on skin flora of the abdominal and inguinal regions of human subjects as measured by change in microbial flora relative to baseline.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of any race
* Subjects in good general health
* Minimum skin flora baseline requirements on abdomen and groin

Exclusion Criteria:

* Any tattoos, scars, breaks in the skin, or any form of dermatitis, or other skin disorders (including acne) on the applicable test areas
* Topical antimicrobial exposure within 14 days prior to screening and treatment days
* Use of systemic or topical antibiotics, steroid medications, or any other products known to affect the normal microbial flora of the skin within 14 days prior to screening and treatment days

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-03; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad H Bashir, MD, CCRP, Principal Investigator — MicroBioTest Inc.
Locations (1):
- MicroBioTest, Sterling, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a randomized, paired-comparisons design where each subject will receive two of the planned treatments, one on the left side of body and one on the right.
  Each subject provided two abdomen test sites, left or right, and/or two inguinal test sites, left or right. A total of 25 subjects were randomized to the abdomen region and 23 subjects were randomized to the inguinal region resulting in 27 subjects providing 96 application test sites on two anatomical regions.
Units Other Than Participants: Test sites on skin
Groups:
- 3M CHG/IPA - Abdominal Region: Experimental CHG/IPA Prep was randomly assigned to the left or right side of the abdominal test site
- Normal Saline - Abdominal Region: Saline control was randomly assigned to the left or right side of the abdominal test site
- 3M CHG/IPA Prep - Inguinal Region: Experimental CHG/IPA Prep was randomly assigned to the left or right side of the inguinal test site
- Normal Saline - Inguinal Region: Saline control was randomly assigned to the left or right side of the inguinal test site
Period: Overall Study
Arm/Group | 3M CHG/IPA - Abdominal Region | Normal Saline - Abdominal Region | 3M CHG/IPA Prep - Inguinal Region | Normal Saline - Inguinal Region
Started | 25; 25 Test sites on skin | 25; 25 Test sites on skin | 23; 23 Test sites on skin | 23; 23 Test sites on skin
Completed | 19; 19 Test sites on skin | 19; 19 Test sites on skin | 21; 21 Test sites on skin | 21; 21 Test sites on skin
Not Completed | 6; 6 Test sites on skin | 6; 6 Test sites on skin | 2; 2 Test sites on skin | 2; 2 Test sites on skin
Not completed — Did not meet treatment day baseline. | 6 | 5 | 2 | 2
Not completed — Dressing was compromised | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Subjects with average treatment day baseline counts of > or equal to 3.00 log10 CFU/cm2 bilaterally on abdominal (abd) region and/or > or equal to 5.00 log10 CFU/cm2 bilaterally on inguinal (ing) region were included in the analysis.
  27 unique subjects provided 50 abd baseline test sites (25 rt & 25 lt) & 46 ing test sites (23 right & 23 left).
  21 unique subjects provided abd & ing test sites; 4 unique subjects provided abd only test sites; 2 unique subjects provided ing only test sites.
Units Other Than Participants: Test sites on skin
Groups:
- 3M CHG/IPA - Abdominal Region - Left or Right: Experimental CHG/IPA Prep was randomly assigned to the left or right side of the abdominal test site
- Normal Saline - Abdominal Region - Left or Right: Saline control was randomly assigned to the left or right side of the abdominal test site
- 3M CHG/IPA Prep - Inguinal Region - Left or Right: Experimental CHG/IPA Prep was randomly assigned to the left or right side of the inguinal test site
- Normal Saline - Inguinal Region - Left or Right: Saline control was randomly assigned to the left or right side of the inguinal test site
- Total: Total of all reporting groups
Arm/Group | 3M CHG/IPA - Abdominal Region - Left or Right | Normal Saline - Abdominal Region - Left or Right | 3M CHG/IPA Prep - Inguinal Region - Left or Right | Normal Saline - Inguinal Region - Left or Right | Total
Number analyzed (Participants) | 25 | 25 | 23 | 23 | 27
Number analyzed (Test sites on skin) | 25 | 25 | 23 | 23 | 96
Age, Customized [Number; unit: Test sites on skin] — Population: Twenty-seven (27) unique subjects provided 50 abdominal baseline test sites (25 right and 25 left) and 46 inguinal test sites (23 right and 23 left).
  Test sites on skin
    Between 18 and 65 years | 22 | 22 | 20 | 20 | 84
    >=66 years | 3 | 3 | 3 | 3 | 12
Sex/Gender, Customized [Number; unit: Test sites on skin] — Population: Twenty-seven (27) unique subjects provided 50 abdominal baseline test sites (25 right and 25 left) and 46 inguinal test sites (23 right and 23 left).
  Test sites on skin
    Female | 5 | 5 | 3 | 3 | 16
    Male | 20 | 20 | 20 | 20 | 80
Race/Ethnicity, Customized [Number; unit: Test sites on skin] — Population: Twenty-seven (27) unique subjects provided 50 abdominal baseline test sites (25 right and 25 left) and 46 inguinal test sites (23 right and 23 left).
  Test sites on skin
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
    Asian | 12 | 12 | 11 | 11 | 46
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
    Black or African American | 3 | 3 | 4 | 4 | 14
    White | 10 | 10 | 8 | 8 | 36
    More than one race | 0 | 0 | 0 | 0 | 0
    Unknown or not reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — Population: Twenty-seven (27) unique subjects provided 50 abdominal baseline test sites (25 right and 25 left) and 46 inguinal test sites (23 right and 23 left).
  participants
    United States | 25 | 25 | 23 | 23 | 27

OUTCOME MEASURES:

1. Primary Outcome: Measurement of Skin Flora Recovery Post-prep Application Relative to Baseline
Description: The primary measure of persistence is the suppression of regrowth recovery relative to baseline (log10 CFU/cm^2) of skin flora at two defined post-prep sampling times relative to baseline.
Time Frame: Baseline, 48 hours and 72 hours post-prep application
Population: Number analyzed includes subjects who met baseline requirements
Measure: Mean (Standard Deviation); unit: Log10 CFU/cm^2
Groups:
- 3M CHG/IPA Prep - Abdominal Region: Experimental CHG/IPA Prep was randomly assigned to the left or right side of the abdominal test site
Arm/Group | Normal Saline - Abdominal Region | 3M CHG/IPA Prep - Abdominal Region | Normal Saline - Inguinal Region | 3M CHG/IPA Prep - Inguinal Region
Number analyzed (Participants) | 20 | 19 | 21 | 21
Log10 CFU/cm^2
  48-hour timepoint | 0.91 (0.78) | 2.81 (0.97) | 0.59 (0.79) | 2.96 (1.07)
  72-hour timepoint: number analyzed (Participants) | 19 | 19 | 21 | 21
  72-hour timepoint | 0.93 (1.07) | 2.44 (1.34) | 0.51 (0.73) | 2.91 (1.60)
Statistical Analysis 1: Comparison: Normal Saline - Abdominal Region vs 3M CHG/IPA Prep - Abdominal Region; 48 hours post treatment time point. The primary analysis used a modified intent to treat population. Subjects were excluded who did not meet the treatment day baseline requirement of greater than or equal to 3.0 log10 CFU/cm^2 on the abdomen. The null hypothesis is that there is no difference in log10 CFU/cm^2 recovery between arms; Test type: Superiority; p < 0.0001, Paired t-test; Mean Difference (Final Values) = 1.97, 95% CI 2-sided [0.51 to 4.10], Standard Error of Mean 0.24
Statistical Analysis 2: Comparison: Normal Saline - Inguinal Region vs 3M CHG/IPA Prep - Inguinal Region; 48 hours post treatment. The primary analysis used a modified intent to treat population. Subjects were excluded who did not meet the treatment day baseline requirement of greater than or equal to 3.0 log10 CFU/cm^2 on the groin. The null hypothesis is that there is no difference in log10 CFU/cm^2 recovery between arms; Test type: Superiority; p = 0.0001, Paired t-test; Mean Difference (Final Values) = 2.37, 95% CI 2-sided [0.60 to 5.75], Standard Error of Mean 0.29
Statistical Analysis 3: Comparison: Normal Saline - Abdominal Region vs 3M CHG/IPA Prep - Abdominal Region; 72 hours post treatment. The primary analysis used a modified intent to treat population. Subjects were excluded who did not meet the treatment day baseline requirement of greater than or equal to 3.0 log10 CFUcm2 on the groin. The null hypothesis is that there is no difference in log10 CFU/cm^2 recovery between arms; Test type: Superiority; p = 0.0001, Paired t-test; Mean Difference (Final Values) = 1.51, 95% CI 2-sided [0.17 to 3.75], Standard Error of Mean 0.23
Statistical Analysis 4: Comparison: Normal Saline - Inguinal Region vs 3M CHG/IPA Prep - Inguinal Region; [analysis description as in outcome 1, analysis 3]; Test type: Superiority; p = 0.0001, Paired t-test; Mean Difference (Final Values) = 2.40, 95% CI 2-sided [0.13 to 5.04], Standard Error of Mean 0.33

2. Secondary Outcome: Safety as Assessed by Skin Irritation Scores Coded by Study Staff
Description: For the conditions of erythema, edema, rash, and dryness, a rating of 0 (no reaction), 1 (mild and/or transient, limited to sensitive area), 2 (moderate, persisting over much of the product-exposed area), or 3 (severe, extending over most or all of the product-exposed area) was recorded on the Skin Irritation Rating form of the eCRF.
Time Frame: 48 hours and 72 hours post-product application
Population: Data from the 48-hour and 72-hour timepoints were combined for each skin condition category of erythema, edema, rash and erythema since all ratings for all subjects at all timepoints were scored as zero (no reaction) for all subjects.
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- 3M CHG/IPA - Abdominal Area; 3M CHG/IPA - Inguinal Area: Chlorhexidine (CHG) 2% / Isopropyl alcohol (IPA) 70%
  3M CHG/IPA Surgical Skin Preparation: Chlorhexidine gluconate 2% / Isopropyl alcohol 70%
- Normal Saline - Abdominal Area; Normal Saline - Inguinal Area: 0.9% sodium chloride with applicator
  Normal Saline: 0.9% sodium chloride applied with foam applicator
Arm/Group | 3M CHG/IPA - Abdominal Area | Normal Saline - Abdominal Area | 3M CHG/IPA - Inguinal Area | Normal Saline - Inguinal Area
Number analyzed (Participants) | 25 | 25 | 23 | 23
Score on a scale
  Erythema: 48-hour timepoint | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Erythema: 72-hour timepoint | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Edema: 48-hour timepoint | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Edema: 72-hour timepoint | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Rash: 48-hour timepoint | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Rash: 72-hour timepoint | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Dryness: 48-hour timepoint | 0 (0) | 0 (0) | 0 (0) | 0 (0)
  Dryness: 72-hour timepoint | 0 (0) | 0 (0) | 0 (0) | 0 (0)

3. Secondary Outcome: Safety as Assessed by Adverse Events
Description: Number of subjects with adverse events as self-reported or identified by study staff
Time Frame: To 72 hours post treatment
Population: Adverse event reports through the treatment period, that is both 48 and 72 hours post dose.
Measure: Count of Participants; unit: Participants
Groups:
- 3M CHG/IPA - Abdomen: Chlorhexidine (CHG) 2% / Isopropyl alcohol (IPA) 70%
  3M CHG/IPA Surgical Skin Preparation: Chlorhexidine gluconate 2% / Isopropyl alcohol 70%
  Applied to the abdominal area
- Normal Saline - Abdomen: 0.9% sodium chloride with applicator
  Normal Saline: 0.9% sodium chloride applied with foam applicator
  Applied to the abdominal area
- 3M CHG/IPA - Inguinal: Chlorhexidine (CHG) 2% / Isopropyl alcohol (IPA) 70%
  3M CHG/IPA Surgical Skin Preparation: Chlorhexidine gluconate 2% / Isopropyl alcohol 70%
  Applied to the inguinal area
- Normal Saline - Inguinal: 0.9% sodium chloride with applicator
  Normal Saline: 0.9% sodium chloride applied with foam applicator
  Applied to the inguinal area
Arm/Group | 3M CHG/IPA - Abdomen | Normal Saline - Abdomen | 3M CHG/IPA - Inguinal | Normal Saline - Inguinal
Number analyzed (Participants) | 25 | 25 | 23 | 23
Participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the treatment phase of the study. The product remained on the skin for approximately 72 hours post.
Arm/Group | 3M CHG/IPA - Abdomen | Normal Saline - Abdomen | 3M CHG/IPA - Inguinal | Normal Saline - Inguinal
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25 | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/23 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No